CLINICAL TRIAL: NCT01111591
Title: Prospective, Randomized, Open-label, Controlled Trial of Cyclooxygenase-2 Inhibitor (Celecoxib; Celebrex®) for Adjuvant Anticancer Effect in Patients With Biliary-pancreas Cancer.
Brief Title: Cyclooxygenase-2 Inhibitor for Adjuvant Anticancer Effect in Patients With Biliary-pancreas Cancer
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Seoul National University Hospital (Other)
Collaborators: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Ho-Seong Han, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SNUBH-GS-HBP2; B-0712-052-006 (local IRB) (Other: Seoul National University Bundang Hospital)
Record Dates: First submitted 2009-03-31; First posted 2010-04-27 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Bile Duct Cancer; Pancreatic Cancer
Keywords: Cyclooxygenase-2 inhibitor (Celecoxib); Extrahepatic bile duct cancer; Pancreas cancer
MeSH Terms: conditions — Bile Duct Neoplasms; Pancreatic Neoplasms | interventions — Cyclooxygenase 2 Inhibitors; Celecoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 2. Bile duct cancer - control (No Intervention): Bile duct cancer patients do not administration of COX inhibitor
- 3. Pancreas cancer - experimental (Experimental): Pancreas cancer patients take a COX2 inhibitor 200mg every 12hours for 6 months
  Interventions: Drug: Cox2 inhibitor (Celecoxib)
- 4. Pancreas cancer - control (No Intervention): Pancreas cancer patients do not administration of COX inhibitor
- Bile duct cancer - experimental (Experimental): Bile duct cancer patients take a COX2 inhibitor 200mg every 12hours for 6 months
  Interventions: Drug: Cox2 inhibitor (Celecoxib)

INTERVENTIONS:
Drug: Cox2 inhibitor (Celecoxib) — From postoperative third day, administration will be started celecoxib 200mg bid for 6 months for administration group.
  Other Names: Celebrex
  Arms: 3. Pancreas cancer - experimental; Bile duct cancer - experimental

SUMMARY:
In extrahepatic bile duct cancer and pancreatic cancer, we will treat postoperatively with COX2 inhibitor and assess survival rate and recurrent rate.

DETAILED DESCRIPTION:
Patients : total 220 patients

* Extrahepatic bile duct cancer : 55 patients for administration of COX2 55 patients for control group
* Pancreas cancer : 55 patients for administration of COX2 55 patients for control group

Indication

* After operation of extrahepatic bile duct cancer or pancreas cancer
* Age : 19 - 70 years old
* The patients who agree to consent sheet.

Contraindication

* Impossible of administration due to severe postoperative morbidities (bleeding, bowel obstruction, pancreatic fistula, biliary fistula)
* Preexisting heart disease: Ischemic heart disease, Heart failure. Severe uncontrolled hypertension (systolic BP>160)
* Renal insufficiency: CCR < 50 or serum creatinin >3.0
* Hepatic insufficiency: Liver cirrhosis or active hepatitis
* Preexisting allergic reaction history for NSAIDs or Sulfonamide
* Current drug intake: Warfarin. Lithium, Fluconazole, Aspirin, Celecoxib
* Preexisting Asthma. Especially aspirin-sensitive asthma.
* Contraindications to aspirin, clopidogrel or celecoxib
* The patients who refuse trial
* The patients who has Psychogenic problem

Allocation

* We will allocate patients randomly, to administration group or control group

Methods

* From postoperative third day, administration will be started
* celecoxib 200mg bid for 6 months for administration group
* Follow up and assess recurrence rate and survival rate

ELIGIBILITY:
Inclusion Criteria:

* The patients who underwent operation for extrahepatic bile duct cancer or pancreas cancer
* Between 19 and 70 years old
* Agreed to consent sheet

Exclusion Criteria:

* The patients cannot administration of drug due to severe postoperative morbidities.
* Preexisting heart disease: Ischemic heart disease, Heart failure. Severe uncontrolled hypertension (systolic BP>160)
* Renal insufficiency: CCR < 50 or serum creatinin >3.0
* Hepatic insufficiency: Liver cirrhosis or active hepatitis
* Preexisting allergic reaction history for NSAIDs or Sulfonamide
* Current drug intake: Warfarin. Lithium, Fluconazole, Aspirin, Celecoxib
* Preexisting Asthma. Especially aspirin-sensitive asthma.
* Contraindications to aspirin, clopidogrel or celecoxib
* When patients refused
* Patients has psychological problem

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2008-11; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Short term outcome | 2 years
  Recurrent rate and survival rate

SECONDARY OUTCOMES:
Long term outcome | 4 years
  Recurrent rate and survival rate

CONTACTS AND LOCATIONS:
Overall Officials: Ho-Seong Han, Professor, Study Chair — General surgery department
Locations (1):
- Ho-Seong Han, Seonnam City, Gyeon Gi Do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Koo BK, Kim YS, Park KW, Yang HM, Kwon DA, Chung JW, Hahn JY, Lee HY, Park JS, Kang HJ, Cho YS, Youn TJ, Chung WY, Chae IH, Choi DJ, Oh BH, Park YB, Kim HS. Effect of celecoxib on restenosis after coronary angioplasty with a Taxus stent (COREA-TAXUS trial): an open-label randomised controlled study. Lancet. 2007 Aug 18;370(9587):567-74. doi: 10.1016/S0140-6736(07)61295-1. PMID 17707751